CLINICAL TRIAL: NCT04801472
Title: Optimisation of Potential Dental Implant Sites Protection for Rehabilitation in Patients With Head and Neck Cancer: Impact of Virtual Implants Visualisation on Dosimetry (OPPIDOM)
Acronym: OPPIDOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: organisationnal reason
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: Hôpitaux Universitaires de Strasbourg (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-013
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma
Keywords: Radiotherapy; Head and Neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with oral cavity or oropharyngeal squamous cell carcinoma (Other)
  Interventions: Other: Optimisation of dental implant sites protection from irradiation

INTERVENTIONS:
Other: Optimisation of dental implant sites protection from irradiation — Optimal treatment plan validation after two dosimetric computer-tomography scans (with or without radiological guide) and visualisation of virtual dental implants on scanner images.
  Evaluation of toxicity, quality of life and dental implant survival rate

SUMMARY:
This is a monocentric, non-randomized, prospective, in silico feasibility study conducted by Strasbourg Europe Cancerology Institute. The purpose of this study is to evaluate the optimisation of potential dental implant sites protection, without degrading tumor volume coverage, through designation of potential dental implant sites before volume delineation and dosimetry calculations in patients with oropharyngeal or oral cavity squamous cell carcinoma treated by radiotherapy.

DETAILED DESCRIPTION:
35 patients will be included in this study and will benefit from a dental consultation for dental rehabilitation plan elaboration and radiological guide confection. Two dosimetric computer-tomography scans, with or without radiological guide, will be conducted. Virtual dental implants will be visualised by the dental surgeon on scanner images (with or without radiologic guide). After volume delineation and dosimetry calculations, the optimal treatment plan will be validated. Patients will be followed throughout radiotherapy and during 18 months following the end of radiotherapy for evaluation of toxicity, quality of life and dental implant survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old
* Performance Status 0 to 2
* Histologically-confirmed diagnosis of : infiltrating squamous cell carcinoma of the oral cavity or oropharynx
* Indication for an exclusive radiotherapy or post-surgery radiotherapy, with or without chemotherapy
* Indication for a radiotherapy of lymph node areas
* Partial or complete toothlessness requiring rehabilitation
* Signed informed consent from the patient

Exclusion Criteria:

* History of head and neck radiotherapy
* Partial mandibulectomy
* Retarded wound healing or trismus impairing radiological guide preparation
* Patient refusing the study
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Identification of optimal scanner allowing to obtain the greater number of patients with every designated implant sites that are protected | At baseline
  Condition of dental implant sites protection (i.e. with minimal implantation risk, Dmax < 40 Gy), without degrading the coverage of planned targeted volume (≥ 95% of volume receiving 95 % of prescribed dose)

SECONDARY OUTCOMES:
Acute toxicity evaluation | every weeks during radiotherapy
  according to CTCAE v5.0 criteria
Retarded toxicity evaluation | 3 months, 6 months, 12 months, 18 months after the end of radiotherapy
  according to CTCAE v5.0 criteria
Quality of life assessed by the EORTC QLQ-C30 questionnaire | At baseline, every weeks during radiotherapy and at 3 months, 6 months, 12 months, 18 months after the end of radiotherapy
  Score based on 30 items from EORTC QLQ-C30 questionnaire
Quality of life for patient with Head and Neck Cancer assessed by the EORTC QLQ-H&N35 supplementary questionnaire module | At baseline, every weeks during radiotherapy and at 3 months, 6 months, 12 months, 18 months after the end of radiotherapy
  Score based on 35 items from EORTC QLQ-H&N35 questionnaire
Oral health-related impact on patients quality of life assessed by the OHIP-14 questionnaire | At baseline, every weeks during radiotherapy and at 3 months, 6 months, 12 months, 18 months after the end of radiotherapy
  Score based on 14 items from OHIP-14 questionnaire
Implant survival rate | at 3 months, 6 months, 12 months, 18 months after the end of radiotherapy
  Number of implant failure (Albrektsson modified criteria)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France